CLINICAL TRIAL: NCT02592642
Title: Self-Management to Improve Walking Ability in Degenerative Lumbar Spinal Stenosis: the Evaluation of Four Novel Strategies.
Brief Title: the Evaluation of Four Non-operative Treatments for Degenerative Lumbar Spinal Stenosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mount Sinai Hospital, Canada (Other)
Collaborators: The Arthritis Society, Canada (Other)
Responsible Party: Principal Investigator, Carlo Ammendolia, Associate Scientist, Mount Sinai Hospital, Canada
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SOG-13-003
Record Dates: First submitted 2015-10-27; First posted 2015-10-30 (Estimated); Last update posted 2017-08-30 (Actual); Status verified 2017-08

CONDITIONS: Degenerative Lumbar Spinal Stenosis
Keywords: lumbar spinal stenosis; neurogenic claudication; non-operative; treatment; outcomes; clinical trial
MeSH Terms: conditions — Spinal Stenosis | interventions — Self-Management; Videotape Recording

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (6):
- Group 1 (Experimental): Self-management Program, Workbook, Video, Pedometer
  Interventions: Behavioral: Self-management Program, Workbook, Video, Pedometer
- Group 2 (Active Comparator): Instructional Workbook, Video, and Pedometer
  Interventions: Behavioral: Instructional Workbook, Video, and Pedometer
- Group a (Experimental): Para-spinal TENS
  Interventions: Device: Para-spinal TENS
- Group b (Placebo Comparator): Para-spinal Placebo TENS
  Interventions: Device: Para-spinal Placebo TENS
- Group c (Experimental): Prototype Spinal Stenosis Belt
  Interventions: Device: Prototype Spinal Stenosis Belt
- Group d (Sham Comparator): Sham spinal stenosis belt
  Interventions: Device: Sham Spinal Stenosis Belt

INTERVENTIONS:
Behavioral: Self-management Program, Workbook, Video, Pedometer — Participants will attend 12 sessions over a six week period. The following therapies will be provided by licensed chiropractors: instruction on self-management strategies, cognitive behavioural techniques; exercise instruction, manual therapy. An instructional workbook and video will provide education and instruction on how to perform exercises, and reinforce instructions received during the sessions. An exercise diary will outline the frequency and intensity of the exercises. All exercises will be performed twice per day at home with the number, intensity, and frequency increasing weekly. Participants will receive a pedometer and record the maximum number of continuous walking steps and time (minutes) to stop walking due to neurogenic symptoms weekly.
  Arms: Group 1
Behavioral: Instructional Workbook, Video, and Pedometer — Participants will attend one session with a chiropractor at the beginning of the six week treatment period. The chiropractor will provide and explain the instructional workbook and video. The workbook and video will provide education and instruction on how to perform exercises all aimed at improving overall fitness in the back and lower extremity and facilitate lumbar flexion. An exercise diary will outline the frequency and intensity of the exercises. All exercises will be performed twice per day at home with the number, intensity, and frequency increasing weekly. Participants will receive a pedometer and record the maximum number of continuous walking steps and time (minutes) to stop walking due to neurogenic symptoms weekly.
  Arms: Group 2
Device: Para-spinal TENS — Participants randomized to this subgroup will have disposable self-adhesive electrical pads (Blue Sensor P, Ambu A/S, Denmark) applied over the para-spinal musculature from L3 to S1 by a licensed chiropractor. The electrical pad electrodes will be connected to a TENS machine (NeuroTrac TENS from Verity Medical Ltd U.K.) which will be worn by the subject concealed within a waist pouch. The TENS will be programmed for a frequency of 65-100 Hz modulated over 3-second intervals with a pulse width of 100-200 usec, and turned on 2 minutes before the start and during the SPWT. Current intensity will be set to the level of comfort of the patient, approximately 3 milliamps in pilot experiments, and below the level causing muscle twitch.
  Arms: Group a
Device: Para-spinal Placebo TENS — Group b: Participants randomized to this subgroup will have disposable self-adhesive electrical pads (Blue Sensor P, Ambu A/S, Denmark) applied over the para-spinal muscular from L3 to S1 by a licensed chiropractor. The electrical pad electrodes will be connected to a TENS machine [NeuroTrac TENS from Verity Medical Ltd (U.K.)] which will be worn by the subject concealed within a waist pouch. The TENS will be programmed using a transient placebo frequency and intensity (45) i.e. the unit will be active for the first 30 seconds then ramping down to zero stimulus over 15 seconds and worn from 2 minutes before the start and during the Self-Paced Walk Test (SPWT).
  Arms: Group b
Device: Prototype Spinal Stenosis Belt — Participants randomized to this subgroup will be fitted with the prototype spinal stenosis belt by a licensed chiropractor. The belt is designed as garment that will snugly fit over the sacrum and pelvic girdle with a pump that place pressure over the sacrum aimed at reducing lordosis.
  Arms: Group c
Device: Sham Spinal Stenosis Belt — Participants randomized to this subgroup will have a standard lumbar support belt (Tensor Adjustable Back Brace from 3M, 207744) fitted around the lumbar spine above the iliac crest comfortably according the manufacturer's instructions for wear. We speculate that the placement of the stenosis belt around the lumbar spine should not have any impact on the lumbar lordosis.
  Arms: Group d

SUMMARY:
Arthritis of the spine causes narrowing of the spinal canals and compression of the spinal nerves traveling into the legs, limiting walking ability. The vast majority of individuals with arthritis of the spine are not suited for surgery and most receive non-surgical treatment. However, we do not know what non-surgical treatments are effective in improving walking in these people. The purpose of our research is to test four new treatments for arthritis of the spine to see if they can improve walking ability. Each treatment approach focuses on the changes that occur in the spine and the whole person as a result of the arthritis that directly or indirectly impacts the ability to walk and perform usual daily activities. Because arthritis of the spine is a chronic condition usually does not go away, it is important that people acquire the knowledge, skills, and tools to manage their condition on their own. The treatments that investigators plan to test as part of this research proposal are aimed at achieving this goal. However, before the investigators can promote the use of these treatments they need to formally test them using strict scientific methods to make sure they do more good than harm. The four treatments include 1) a six week training program referred to as "Boot Camp for Stenosis" which provides one-on-one training on exercise and self-management strategies 2) a patient educational workbook and video on how to self-manage, 3) an electrical device that is placed on the lower back to reduce nerve pain when walking and 4) a spinal stenosis belt that people can wear to reduce pressure on the nerves while walking. The plan is to assess the change in walking distance using the various treatments and assess what impact the treatments have on peoples' overall function and quality of life. Innovative treatment approaches with a long term perspective are urgently needed to deal with the growing number of people with arthritis of the spine who are disabled. It is likely that there is not one solution to this problem - many people will require more than one type of treatment, but an important first step is to determine which treatments are effective, then tailor the treatments to the needs of each person.

DETAILED DESCRIPTION:
Degenerative lumbar spinal stenosis (DLSS) or osteoarthritis of the spine is a leading cause of pain, disability, and loss of independence in older adults. It is a chronic disease caused by age related degenerative narrowing (stenosis) of the spinal canal that can lead to compression and ischemia of the spinal nerves (neuro-ischemia). The clinical syndrome of DLSS is known as neurogenic claudication. It is characterized by bilateral or unilateral buttock and/or lower extremity pain, heaviness, numbness, tingling or weakness, precipitated by walking and standing and relieved by sitting and bending forward. Limited walking ability is the dominant functional impairment caused by DLSS. Those afflicted have greater walking limitations than individuals with knee or hip osteoarthritis and greater functional limitations than those with congestive heart failure, chronic obstructive lung disease or systemic lupus erythematosus. Inability to walk among individuals with DLSS leads to a sedentary lifestyle and a progressive decline in health status. The prevalence and economic burden of DLSS is growing exponentially due to the aging population. Although DLSS is the most common reason for spine surgery in individuals over the age of 65, only very few DLSS patients receive surgery. The vast majority of individuals with DLSS receive non-surgical care. However, what constitutes effective non-surgical care is unknown. Self-management strategies may be a practical and effective means to improve walking ability, functional status, and quality of life in this chronic arthritic and often progressive condition. The investigators have conducted two systematic reviews of the literature, one assessing the effectiveness of non-surgical treatments for neurogenic claudication which included randomized controlled trials (RCTs) assessing improvements in pain, disability, quality of life or global improvement; the other evaluated the effectiveness of surgical or non-surgical interventions and included only RCTs that assessed improved walking ability. the investigators learned from these reviews that the evidence for interventions that improve outcomes including walking ability in neurogenic claudication due to DLSS is lacking. The evidence published thus far on this topic has been of low or of very low quality, prohibiting the formulation of evidence-based recommendations for clinical practice. Moreover, the investigators identified no RCTs that examined a self-management approach to the treatment of DLSS.

In addition to the structural arthritic changes causing narrowing of the spinal canal, DLSS has an important dynamic component. The volume of the spinal canal and degree of epidural pressure and ischemia of the spinal nerves can change depending on spinal posture. Both lumbar flexion (stooping forward), and sitting increase the diameter of the canal and reduce spinal nerve ischemia, and correspond with a reduction or elimination of lower extremity symptoms. Conversely, lumbar extension or increasing the lumbar lordosis (which occurs when standing) reduces the diameter of the spinal canal and increases spinal nerve ischemia, and corresponds with increased lower extremity symptoms. The ability to reduce symptoms of DLSS by changing spinal posture/structural alignment and/or increasing blood flow to the spinal nerve provides potential mechanisms for developing interventions to improve symptoms and walking ability.

First, the investigators have designed and implemented a novel six week self-management training program for DLSS over the past 3 years at the Spinal Stenosis Clinic at the Rebecca MacDonald Centre for Arthritis and Auto-immune Diseases at Mount Sinai Hospital (MSH). The goal of the training program is to provide patients with the knowledge, skills, self-confidence, and physical capacity to manage their symptoms and maximize their function. The program is multi-modal, tailored and directed to the structural, functional, physiological and psychosocial consequences of DLSS. Particular emphasis is placed on exercise instruction to build core and lower extremity strength and enable individuals to achieve optimal posture during standing and walking.

There are numerous human studies demonstrating significant reduction in laboratory induced ischemic pain in the lower and upper extremities with paraspinal TENS compared to placebo TENS. Moreover, there is low quality evidence from one case series suggesting that electrical stimulation may be effective for the management of neurogenic claudication. Higher quality studies are needed to assess whether paraspinal TENS applied while walking improves walking ability, as this could be an innovative, convenient, and inexpensive self-management strategy for DLSS patients.

Finally, the investigators have designed a prototype spinal stenosis belt with the Ontario College of Art and Design. The belt is designed as garment that will snugly fit over the sacrum and pelvic girdle with a pump that place pressure over the sacrum with the aim to reduce the lumbar lordosis and maximize the spinal canal diameter when walking. The investigators hypothesize the belt will reduce the lumbar lordosis and alleviate epidural pressure and neuro-ischemia while standing and walking. The investigators identified two preliminary studies evaluating back belts, supports or braces for DLSS, none of which were RCTs. These studies found significant improvements in walking distance with the use of a back corset; however both studies had a high risk of bias.

OBJECTIVES AND HYPOTHESES The overall goal of this study is to assess the effectiveness of four self-management strategies in improving walking ability among patients with DLSS. The investigators primary objective is to compare the effectiveness of a comprehensive six week self-management training program that includes a patient instructional workbook, video and pedometer to a patient workbook, video and pedometer alone. The investigators secondary objectives are: 1) to compare the change in walking capacity from baseline when using superficially applied para-spinal TENS versus placebo para-spinal TENS applied during walking and 2) to compare the change in walking capacity from baseline while wearing a novel spinal stenosis belt to the use of a sham spinal stenosis belt while walking. The investigators hypothesize that the self-management training program with workbook, video and pedometer will be more effective in improving walking capacity and functional outcomes than the use of a workbook, video and pedometer alone. Furthermore, the investigators hypothesize that para-spinal TENS or the novel spinal stenosis belt used while walking will be more effective in improving walking capacity than placebo TENS or a sham spinal stenosis belt, respectively.

ELIGIBILITY:
Inclusion Criteria:

* Age greater or equal to 50 years
* Clinical symptoms of back and/or radiating lower limb or buttock pain; fatigue or loss of sensation in the lower limbs aggravated by walking and/or standing and relieved by sitting
* Intermittent or persistent pain without progressive neurological dysfunction
* Duration of symptoms and signs for more than 3 months
* Imaging confirmed spinal canal narrowing using MRI, CT scan, myelography or ultrasound
* Clinical signs and symptoms corresponding to segmental level of narrowing identified by imaging
* Patients with degenerative spondylolisthesis are included
* Not considered to be a surgical candidate (in the next 12 months) or patient unwilling to have surgery
* Able to perform mild-moderate exercise
* Able to walk without assistive devices for at least 20 metres and less than 30 minutes continuously
* Able to give written informed consent and complete interviews and questionnaires in English.

Exclusion Criteria:

* Severe degenerative stenosis with intractable pain and progressive neurological dysfunction
* Lumbar spinal stenosis not caused by degeneration
* Lumbar herniated disc diagnosed during the last 12 months
* Previous back surgery for lumbar spinal stenosis or instability
* Underlying spinal disorder such as ankylosing spondylitis, neoplasm, infection or metabolic disease
* Intermittent claudication due to vascular disease
* Severe osteoarthrosis or arthritis of lower extremities causing limited walking ability
* Neurologic disease causing impaired function of the lower limbs, including diabetes
* Psychiatric disorders and /or cognitively impaired

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104 (Actual)
Dates: Start 2014-09; Primary Completion 2017-02-15 (Actual); Study Completion 2017-03-01 (Actual)

PRIMARY OUTCOMES:
Change in The Self-Paced Walk Test | Change from baseline to 6 weeks (immediately post-intervention), 3 months, 6 months, and 12 months post-intervention
  The Self-Paced Walk Test requires subjects to walk on a level surface without support at their own pace until forced to stop due to symptoms of DLSS or after a time limit of 30 minutes (54). Test termination will be defined as a complete stop of 3 seconds. A blinded assessor will follow one meter behind the subject, without conversing, with a distance instrument (Lufkin Pro-Series Model PSMW38), and stop watch. Distance walked and time to test termination will be recorded.

SECONDARY OUTCOMES:
Zurich Claudication Questionnaire | change from baseline to 6 weeks (immediately post-intervention), 3 months, 6 months, and 12 months post-intervention
  The Zurich Claudication Questionnaire (ZCQ), also known as the Swiss Spinal Stenosis Scale, will be used as a measure of physical function and symptom severity. The questionnaire consists of three scales; a physical performance scale, a symptom severity scale, and a patient satisfaction scale (56, 57). The physical performance scale consists of five questions related to walking ability. The mean un-weighted score will be calculated. The symptom scale consists of seven questions pertaining to overall severity of pain, pain frequency, back pain and, pain in the leg, numbness, weakness, and balance disturbance.
Oswestry Disability Index | change from baseline to 6 weeks (immediately post-intervention), 3 months, 6 months, and 12 months post-intervention
  The Oswestry Disability Index will be used to assess back related disability. The total score will be calculated where 0 represents no disability and 100 represent the worse possible disability. We will also record separately the score of the walking section (ODI walk) of the ODI.
Numeric Rating Scale | change from baseline to 6 weeks (immediately post-intervention), 3 months, 6 months, and 12 months post-intervention
  The Numeric Rating Scale will be used to assess leg and back pain intensity while walking. It is an 11-point scale anchored by two extremes of pain intensity ranging from 0 (referring to "No pain") to 10 (referring to "Pain as bad as it could be").
Medical Outcomes Study Short-Form Health Survey version two (SF-36) | change form baseline to 6 weeks (immediately post-intervention), 3 months, 6 months, and 12 months post-intervention
  We will use the Medical Outcomes Study Short-Form Health Survey version two (SF-36) to measure health-related quality of life (H-RQoL). The SF-36 has 36 items which measure the H-RQoL of a subject. Two summary scores can be computed: the physical component score and the mental component score.
Centre for Epidemiological Studies Depression Scale | Change from baseline to 6 weeks (immediately post-intervention), 3 months, 6 months, and 12 months post-intervention
  The Center for Epidemiological Studies-Depression Scale (CES-D) will be used to measure depressive symptomatology in the previous week. The CES-D is a widely used 20-item self-report scale designed to measure current level of depressive symptomatology in population-based epidemiologic research (65).

CONTACTS AND LOCATIONS:
Overall Officials: Carlo Ammendolia, PhD, Principal Investigator — MOUNT SINAI HOSPITAL
Locations (1):
- Mount Sinai Hospital, Toronto, Ontario, Canada

REFERENCES:
- [Background] Fanuele JC, Birkmeyer NJ, Abdu WA, Tosteson TD, Weinstein JN. The impact of spinal problems on the health status of patients: have we underestimated the effect? Spine (Phila Pa 1976). 2000 Jun 15;25(12):1509-14. doi: 10.1097/00007632-200006150-00009. PMID 10851099
- [Background] Takahashi K, Kagechika K, Takino T, Matsui T, Miyazaki T, Shima I. Changes in epidural pressure during walking in patients with lumbar spinal stenosis. Spine (Phila Pa 1976). 1995 Dec 15;20(24):2746-9. doi: 10.1097/00007632-199512150-00017. PMID 8747254
- [Background] Diggle P. Analysis of longitudinal data. Press OU, editor. New York2009.
- [Background] Katz JN, Dalgas M, Stucki G, Katz NP, Bayley J, Fossel AH, Chang LC, Lipson SJ. Degenerative lumbar spinal stenosis. Diagnostic value of the history and physical examination. Arthritis Rheum. 1995 Sep;38(9):1236-41. doi: 10.1002/art.1780380910. PMID 7575718
- [Background] Suri P, Rainville J, Kalichman L, Katz JN. Does this older adult with lower extremity pain have the clinical syndrome of lumbar spinal stenosis? JAMA. 2010 Dec 15;304(23):2628-36. doi: 10.1001/jama.2010.1833. PMID 21156951
- [Background] Winter CC, Brandes M, Muller C, Schubert T, Ringling M, Hillmann A, Rosenbaum D, Schulte TL. Walking ability during daily life in patients with osteoarthritis of the knee or the hip and lumbar spinal stenosis: a cross sectional study. BMC Musculoskelet Disord. 2010 Oct 12;11:233. doi: 10.1186/1471-2474-11-233. PMID 20939866
- [Background] Iversen MD, Katz JN. Examination findings and self-reported walking capacity in patients with lumbar spinal stenosis. Phys Ther. 2001 Jul;81(7):1296-306. PMID 11444993
- [Background] Jonsson B, Annertz M, Sjoberg C, Stromqvist B. A prospective and consecutive study of surgically treated lumbar spinal stenosis. Part I: Clinical features related to radiographic findings. Spine (Phila Pa 1976). 1997 Dec 15;22(24):2932-7. doi: 10.1097/00007632-199712150-00016. PMID 9431629
- [Background] Jansson KA, Nemeth G, Granath F, Jonsson B, Blomqvist P. Health-related quality of life (EQ-5D) before and one year after surgery for lumbar spinal stenosis. J Bone Joint Surg Br. 2009 Feb;91(2):210-6. doi: 10.1302/0301-620X.91B2.21119. PMID 19190056
- [Background] Deyo RA, Mirza SK, Martin BI, Kreuter W, Goodman DC, Jarvik JG. Trends, major medical complications, and charges associated with surgery for lumbar spinal stenosis in older adults. JAMA. 2010 Apr 7;303(13):1259-65. doi: 10.1001/jama.2010.338. PMID 20371784
- [Background] Chen E, Tong KB, Laouri M. Surgical treatment patterns among Medicare beneficiaries newly diagnosed with lumbar spinal stenosis. Spine J. 2010 Jul;10(7):588-94. doi: 10.1016/j.spinee.2010.02.026. Epub 2010 Apr 8. PMID 20381431
- [Background] Ammendolia C, Stuber K, de Bruin LK, Furlan AD, Kennedy CA, Rampersaud YR, Steenstra IA, Pennick V. Nonoperative treatment of lumbar spinal stenosis with neurogenic claudication: a systematic review. Spine (Phila Pa 1976). 2012 May 1;37(10):E609-16. doi: 10.1097/BRS.0b013e318240d57d. PMID 22158059
- [Background] Tran DQ, Duong S, Finlayson RJ. Lumbar spinal stenosis: a brief review of the nonsurgical management. Can J Anaesth. 2010 Jul;57(7):694-703. doi: 10.1007/s12630-010-9315-3. Epub 2010 Apr 29. PMID 20428988
- [Background] May S, Comer C. Is surgery more effective than non-surgical treatment for spinal stenosis, and which non-surgical treatment is more effective? A systematic review. Physiotherapy. 2013 Mar;99(1):12-20. doi: 10.1016/j.physio.2011.12.004. Epub 2012 Apr 16. PMID 23219644
- [Background] Atlas SJ, Keller RB, Wu YA, Deyo RA, Singer DE. Long-term outcomes of surgical and nonsurgical management of lumbar spinal stenosis: 8 to 10 year results from the maine lumbar spine study. Spine (Phila Pa 1976). 2005 Apr 15;30(8):936-43. doi: 10.1097/01.brs.0000158953.57966.c0. PMID 15834339
- [Background] Ammendolia C, Stuber K, Tomkins-Lane C, Schneider M, Rampersaud YR, Furlan AD, Kennedy CA. What interventions improve walking ability in neurogenic claudication with lumbar spinal stenosis? A systematic review. Eur Spine J. 2014 Jun;23(6):1282-301. doi: 10.1007/s00586-014-3262-6. Epub 2014 Mar 15. PMID 24633719
- [Background] Tomkins-Lane CC, Battie MC. Validity and reproducibility of self-report measures of walking capacity in lumbar spinal stenosis. Spine (Phila Pa 1976). 2010 Nov 1;35(23):2097-102. doi: 10.1097/BRS.0b013e3181f5e13b. PMID 20938380
- [Background] Iversen MD, Hammond A, Betteridge N. Self-management of rheumatic diseases: state of the art and future perspectives. Ann Rheum Dis. 2010 Jun;69(6):955-63. doi: 10.1136/ard.2010.129270. Epub 2010 May 6. PMID 20448289
- [Background] Warsi A, LaValley MP, Wang PS, Avorn J, Solomon DH. Arthritis self-management education programs: a meta-analysis of the effect on pain and disability. Arthritis Rheum. 2003 Aug;48(8):2207-13. doi: 10.1002/art.11210. PMID 12905474
- [Background] Bodenheimer T, Lorig K, Holman H, Grumbach K. Patient self-management of chronic disease in primary care. JAMA. 2002 Nov 20;288(19):2469-75. doi: 10.1001/jama.288.19.2469. PMID 12435261
- [Background] Oliveira VC, Ferreira PH, Maher CG, Pinto RZ, Refshauge KM, Ferreira ML. Effectiveness of self-management of low back pain: systematic review with meta-analysis. Arthritis Care Res (Hoboken). 2012 Nov;64(11):1739-48. doi: 10.1002/acr.21737. PMID 22623349
- [Background] Chung SS, Lee CS, Kim SH, Chung MW, Ahn JM. Effect of low back posture on the morphology of the spinal canal. Skeletal Radiol. 2000 Apr;29(4):217-23. doi: 10.1007/s002560050596. PMID 10855470
- [Background] Madsen R, Jensen TS, Pope M, Sorensen JS, Bendix T. The effect of body position and axial load on spinal canal morphology: an MRI study of central spinal stenosis. Spine (Phila Pa 1976). 2008 Jan 1;33(1):61-7. doi: 10.1097/BRS.0b013e31815e395f. PMID 18165750
- [Background] Kanno H, Ozawa H, Koizumi Y, Morozumi N, Aizawa T, Kusakabe T, Ishii Y, Itoi E. Dynamic change of dural sac cross-sectional area in axial loaded magnetic resonance imaging correlates with the severity of clinical symptoms in patients with lumbar spinal canal stenosis. Spine (Phila Pa 1976). 2012 Feb 1;37(3):207-13. doi: 10.1097/BRS.0b013e3182134e73. PMID 21301392
- [Background] Takahashi K, Miyazaki T, Takino T, Matsui T, Tomita K. Epidural pressure measurements. Relationship between epidural pressure and posture in patients with lumbar spinal stenosis. Spine (Phila Pa 1976). 1995 Mar 15;20(6):650-3. PMID 7604339
- [Background] Kalichman L, Cole R, Kim DH, Li L, Suri P, Guermazi A, Hunter DJ. Spinal stenosis prevalence and association with symptoms: the Framingham Study. Spine J. 2009 Jul;9(7):545-50. doi: 10.1016/j.spinee.2009.03.005. Epub 2009 Apr 23. PMID 19398386
- [Background] Gempt J, Rothoerl RD, Grams A, Meyer B, Ringel F. Effect of lumbar spinal stenosis and surgical decompression on erectile function. Spine (Phila Pa 1976). 2010 Oct 15;35(22):E1172-7. doi: 10.1097/BRS.0b013e3181e7d98b. PMID 20881655
- [Background] Wood DW, Haig AJ, Yamakawa KS. Fear of movement/(re)injury and activity avoidance in persons with neurogenic versus vascular claudication. Spine J. 2012 Apr;12(4):292-300. doi: 10.1016/j.spinee.2012.02.015. Epub 2012 Apr 4. PMID 22480530
- [Background] Sinikallio S, Aalto T, Airaksinen O, Herno A, Kroger H, Savolainen S, Turunen V, Viinamaki H. Depression and associated factors in patients with lumbar spinal stenosis. Disabil Rehabil. 2006 Apr 15;28(7):415-22. doi: 10.1080/09638280500192462. PMID 16507504
- [Background] Ostelo RW, van Tulder MW, Vlaeyen JW, Linton SJ, Morley SJ, Assendelft WJ. Behavioural treatment for chronic low-back pain. Cochrane Database Syst Rev. 2005 Jan 25;(1):CD002014. doi: 10.1002/14651858.CD002014.pub2. PMID 15674889
- [Background] Linton SJ, Andersson T. Can chronic disability be prevented? A randomized trial of a cognitive-behavior intervention and two forms of information for patients with spinal pain. Spine (Phila Pa 1976). 2000 Nov 1;25(21):2825-31; discussion 2824. doi: 10.1097/00007632-200011010-00017. PMID 11064530
- [Background] Whitman JM, Flynn TW, Childs JD, Wainner RS, Gill HE, Ryder MG, Garber MB, Bennett AC, Fritz JM. A comparison between two physical therapy treatment programs for patients with lumbar spinal stenosis: a randomized clinical trial. Spine (Phila Pa 1976). 2006 Oct 15;31(22):2541-9. doi: 10.1097/01.brs.0000241136.98159.8c. PMID 17047542
- [Background] Whitman JM, Flynn TW, Fritz JM. Nonsurgical management of patients with lumbar spinal stenosis: a literature review and a case series of three patients managed with physical therapy. Phys Med Rehabil Clin N Am. 2003 Feb;14(1):77-101, vi-vii. doi: 10.1016/s1047-9651(02)00076-1. PMID 12622484
- [Background] Murphy DR, Hurwitz EL, Gregory AA, Clary R. A non-surgical approach to the management of lumbar spinal stenosis: a prospective observational cohort study. BMC Musculoskelet Disord. 2006 Feb 23;7:16. doi: 10.1186/1471-2474-7-16. PMID 16504078
- [Background] Woolf CJ. Transcutaneous electrical nerve stimulation and the reaction to experimental pain in human subjects. Pain. 1979 Oct;7(2):115-127. doi: 10.1016/0304-3959(79)90003-4. PMID 523169
- [Background] Foster NE, Baxter F, Walsh DM, Baxter GD, Allen JM. Manipulation of transcutaneous electrical nerve stimulation variables has no effect on two models of experimental pain in humans. Clin J Pain. 1996 Dec;12(4):301-10. doi: 10.1097/00002508-199612000-00009. PMID 8969875
- [Background] Walsh DM, Liggett C, Baxter D, Allen JM. A double-blind investigation of the hypoalgesic effects of transcutaneous electrical nerve stimulation upon experimentally induced ischaemic pain. Pain. 1995 Apr;61(1):39-45. doi: 10.1016/0304-3959(94)00147-7. PMID 7644247
- [Background] Seenan C, Roche PA, Tan CW, Mercer T. Modification of experimental, lower limb ischemic pain with transcutaneous electrical nerve stimulation. Clin J Pain. 2012 Oct;28(8):693-9. doi: 10.1097/AJP.0b013e318242fccb. PMID 22209796
- [Background] Roche PAT, H; Stanton WR. Modification of induced ischaemic pain by placebo electrotherapy. . Physiotherapy Theory Practice. 2002;18:131-9.
- [Background] Inoue M, Hojo T, Nakajima M, Kitakoji H, Itoi M, Katsumi Y. Pudendal nerve electroacupuncture for lumbar spinal canal stenosis - a case series. Acupunct Med. 2008 Sep;26(3):140-4. doi: 10.1136/aim.26.3.140. PMID 18818559
- [Background] Weiss HR, Dallmayer R. Brace treatment of spinal claudication in an adolescent with a grade IV spondylosisthesis--a case report. Stud Health Technol Inform. 2006;123:590-3. PMID 17108493
- [Background] Prateepavanich P, Thanapipatsiri S, Santisatisakul P, Somshevita P, Charoensak T. The effectiveness of lumbosacral corset in symptomatic degenerative lumbar spinal stenosis. J Med Assoc Thai. 2001 Apr;84(4):572-6. PMID 11460971
- [Background] Elashoff J. nQuery Advisor. Version 70 User's Guide. 7.0 User's Guide ed. Los Angeles, CA USA2007.
- [Background] Rakel B, Cooper N, Adams HJ, Messer BR, Frey Law LA, Dannen DR, Miller CA, Polehna AC, Ruggle RC, Vance CG, Walsh DM, Sluka KA. A new transient sham TENS device allows for investigator blinding while delivering a true placebo treatment. J Pain. 2010 Mar;11(3):230-8. doi: 10.1016/j.jpain.2009.07.007. Epub 2009 Nov 27. PMID 19945354
- [Background] Woby SR, Urmston M, Watson PJ. Self-efficacy mediates the relation between pain-related fear and outcome in chronic low back pain patients. Eur J Pain. 2007 Oct;11(7):711-8. doi: 10.1016/j.ejpain.2006.10.009. Epub 2007 Jan 10. PMID 17218132
- [Background] Lorig KR, Sobel DS, Ritter PL, Laurent D, Hobbs M. Effect of a self-management program on patients with chronic disease. Eff Clin Pract. 2001 Nov-Dec;4(6):256-62. PMID 11769298
- [Background] Bodack MP, Monteiro M. Therapeutic exercise in the treatment of patients with lumbar spinal stenosis. Clin Orthop Relat Res. 2001 Mar;(384):144-52. doi: 10.1097/00003086-200103000-00017. PMID 11249159
- [Background] Pua YH, Cai CC, Lim KC. Treadmill walking with body weight support is no more effective than cycling when added to an exercise program for lumbar spinal stenosis: a randomised controlled trial. Aust J Physiother. 2007;53(2):83-9. doi: 10.1016/s0004-9514(07)70040-5. PMID 17535143
- [Background] Ellis RF, Hing WA. Neural mobilization: a systematic review of randomized controlled trials with an analysis of therapeutic efficacy. J Man Manip Ther. 2008;16(1):8-22. doi: 10.1179/106698108790818594. PMID 19119380
- [Background] Maitland G. Peripheral Manipulation. Butterworth-Heinemann O, editor1991.
- [Background] McGill S. Low back disorders: evidence-based prevention and rehabilitation: Human Kinetics 1; 2007.
- [Background] Gudavalli MR, Cambron JA, McGregor M, Jedlicka J, Keenum M, Ghanayem AJ, Patwardhan AG. A randomized clinical trial and subgroup analysis to compare flexion-distraction with active exercise for chronic low back pain. Eur Spine J. 2006 Jul;15(7):1070-82. doi: 10.1007/s00586-005-0021-8. Epub 2005 Dec 8. PMID 16341712
- [Background] Tomkins CC, Battie MC, Rogers T, Jiang H, Petersen S. A criterion measure of walking capacity in lumbar spinal stenosis and its comparison with a treadmill protocol. Spine (Phila Pa 1976). 2009 Oct 15;34(22):2444-9. doi: 10.1097/BRS.0b013e3181b03fc8. PMID 19829259
- [Background] Rainville J, Childs LA, Pena EB, Suri P, Limke JC, Jouve C, Hunter DJ. Quantification of walking ability in subjects with neurogenic claudication from lumbar spinal stenosis--a comparative study. Spine J. 2012 Feb;12(2):101-9. doi: 10.1016/j.spinee.2011.12.006. Epub 2011 Dec 29. PMID 22209240
- [Background] Stucki G, Daltroy L, Liang MH, Lipson SJ, Fossel AH, Katz JN. Measurement properties of a self-administered outcome measure in lumbar spinal stenosis. Spine (Phila Pa 1976). 1996 Apr 1;21(7):796-803. doi: 10.1097/00007632-199604010-00004. PMID 8779009
- [Background] Pratt RK, Fairbank JC, Virr A. The reliability of the Shuttle Walking Test, the Swiss Spinal Stenosis Questionnaire, the Oxford Spinal Stenosis Score, and the Oswestry Disability Index in the assessment of patients with lumbar spinal stenosis. Spine (Phila Pa 1976). 2002 Jan 1;27(1):84-91. doi: 10.1097/00007632-200201010-00020. PMID 11805642
- [Background] Fairbank JC, Couper J, Davies JB, O'Brien JP. The Oswestry low back pain disability questionnaire. Physiotherapy. 1980 Aug;66(8):271-3. No abstract available. PMID 6450426
- [Background] Fritz JM, Irrgang JJ. A comparison of a modified Oswestry Low Back Pain Disability Questionnaire and the Quebec Back Pain Disability Scale. Phys Ther. 2001 Feb;81(2):776-88. doi: 10.1093/ptj/81.2.776. PMID 11175676
- [Background] Wewers ME, Lowe NK. A critical review of visual analogue scales in the measurement of clinical phenomena. Res Nurs Health. 1990 Aug;13(4):227-36. doi: 10.1002/nur.4770130405. PMID 2197679
- [Background] Jensen MP, Karoly P, Braver S. The measurement of clinical pain intensity: a comparison of six methods. Pain. 1986 Oct;27(1):117-126. doi: 10.1016/0304-3959(86)90228-9. PMID 3785962
- [Background] Haley SM, McHorney CA, Ware JE Jr. Evaluation of the MOS SF-36 physical functioning scale (PF-10): I. Unidimensionality and reproducibility of the Rasch item scale. J Clin Epidemiol. 1994 Jun;47(6):671-84. doi: 10.1016/0895-4356(94)90215-1. PMID 7722580
- [Background] Groll DL, To T, Bombardier C, Wright JG. The development of a comorbidity index with physical function as the outcome. J Clin Epidemiol. 2005 Jun;58(6):595-602. doi: 10.1016/j.jclinepi.2004.10.018. PMID 15878473
- [Background] 64. Radloff LS. The CES-D scale A self-report depression scale for research in the general population. Applied psychological measurement. 1977;1(3):385-401
- [Background] Orme JG, Reis J, Herz EJ. Factorial and discriminant validity of the Center for Epidemiological Studies Depression (CES-D) scale. J Clin Psychol. 1986 Jan;42(1):28-33. doi: 10.1002/1097-4679(198601)42:13.0.co;2-t. PMID 3950011
- [Background] Guralnik JM, Simonsick EM, Ferrucci L, Glynn RJ, Berkman LF, Blazer DG, Scherr PA, Wallace RB. A short physical performance battery assessing lower extremity function: association with self-reported disability and prediction of mortality and nursing home admission. J Gerontol. 1994 Mar;49(2):M85-94. doi: 10.1093/geronj/49.2.m85. PMID 8126356
- [Background] Guralnik JM, Ferrucci L, Pieper CF, Leveille SG, Markides KS, Ostir GV, Studenski S, Berkman LF, Wallace RB. Lower extremity function and subsequent disability: consistency across studies, predictive models, and value of gait speed alone compared with the short physical performance battery. J Gerontol A Biol Sci Med Sci. 2000 Apr;55(4):M221-31. doi: 10.1093/gerona/55.4.m221. PMID 10811152
- [Background] Winograd CH, Lemsky CM, Nevitt MC, Nordstrom TM, Stewart AL, Miller CJ, Bloch DA. Development of a physical performance and mobility examination. J Am Geriatr Soc. 1994 Jul;42(7):743-9. doi: 10.1111/j.1532-5415.1994.tb06535.x. PMID 8014350
- [Background] Tinetti ME, Richman D, Powell L. Falls efficacy as a measure of fear of falling. J Gerontol. 1990 Nov;45(6):P239-43. doi: 10.1093/geronj/45.6.p239. PMID 2229948
- [Background] Falls: Assessment and Prevention of Falls in Older People. London: National Institute for Health and Care Excellence (NICE); 2013 Jun. Available from http://www.ncbi.nlm.nih.gov/books/NBK258885/ PMID 25506960
- [Background] Huang TT, Wang WS. Comparison of three established measures of fear of falling in community-dwelling older adults: psychometric testing. Int J Nurs Stud. 2009 Oct;46(10):1313-9. doi: 10.1016/j.ijnurstu.2009.03.010. Epub 2009 Apr 24. PMID 19394017
- [Background] Cohen J. A power primer. Psychol Bull. 1992 Jul;112(1):155-9. doi: 10.1037//0033-2909.112.1.155. PMID 19565683
- [Background] Greenland SR. Introduction to stratified analysis. In Modern Epidemiology. Philadelphia, PA: Lippincott-Raven; 1998.
- [Derived] Ammendolia C, Cote P, Rampersaud YR, Southerst D, Schneider M, Ahmed A, Bombardier C, Hawker G, Budgell B. Effect of active TENS versus de-tuned TENS on walking capacity in patients with lumbar spinal stenosis: a randomized controlled trial. Chiropr Man Therap. 2019 Jun 19;27:24. doi: 10.1186/s12998-019-0245-z. eCollection 2019. PMID 31244992
- [Derived] Ammendolia C, Cote P, Southerst D, Schneider M, Budgell B, Bombardier C, Hawker G, Rampersaud YR. Comprehensive Nonsurgical Treatment Versus Self-directed Care to Improve Walking Ability in Lumbar Spinal Stenosis: A Randomized Trial. Arch Phys Med Rehabil. 2018 Dec;99(12):2408-2419.e2. doi: 10.1016/j.apmr.2018.05.014. Epub 2018 Jun 20. PMID 29935152
- [Derived] Ammendolia C, Cote P, Rampersaud YR, Southerst D, Budgell B, Bombardier C, Hawker G. Effect of TENS Versus Placebo on Walking Capacity in Patients With Lumbar Spinal Stenosis: A Protocol for a Randomized Controlled Trial. J Chiropr Med. 2016 Sep;15(3):197-203. doi: 10.1016/j.jcm.2016.04.001. Epub 2016 Jun 20. PMID 27660596
- [Derived] Ammendolia C, Cote P, Rampersaud YR, Southerst D, Budgell B, Bombardier C, Hawker G. The boot camp program for lumbar spinal stenosis: a protocol for a randomized controlled trial. Chiropr Man Therap. 2016 Jul 18;24:25. doi: 10.1186/s12998-016-0106-y. eCollection 2016. PMID 27433335